CLINICAL TRIAL: NCT00762502
Title: Comparison of Senofilcon A Toric Lenses to Balafilcon A Toric Lenses Over Extended Wear Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR-4498
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2014-11-25 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2015-05

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- senofilcon A toric bilaterally (Active Comparator): senofilcon A lenses worn daily bilaterally (in both eyes) for 3 months, replaced weekly.
  Interventions: Device: senofilcon A toric contact lens
- balafilcon A toric bilaterally (Active Comparator): balafilcon A lenses worn daily bilaterally (in both eyes) for 3 months, replaced weekly.
  Interventions: Device: balafilcon A toric contact lens
- senofilcon A/balafilcon A contralaterally (Active Comparator): senofilcon A lens worn in one eye and balafilcon A lens worn in the other eye (contralaterally), daily for 3 months, replaced weekly.
  Interventions: Device: senofilcon A toric contact lens; Device: balafilcon A toric contact lens

INTERVENTIONS:
Device: senofilcon A toric contact lens — soft contact lens
  Arms: senofilcon A toric bilaterally; senofilcon A/balafilcon A contralaterally
Device: balafilcon A toric contact lens — soft contact lens
  Arms: balafilcon A toric bilaterally; senofilcon A/balafilcon A contralaterally

SUMMARY:
To evaluate two toric contact lenses on the ocular physiology of existing contact lens wearers when used in an extended wear modality of days/six nights.

ELIGIBILITY:
Inclusion Criteria:

* Able to wear study lenses in parameters available
* Non-presbyopes between the ages of 18-45
* Understand and sign informed consent
* Willing to follow the protocol
* Achieve at least 20/30 (6/9) visual acuity (VA) in right eye (OD) and left eye (OS) with study lenses
* Myopia -0.75 to -6.25, cylinder -0.75 to -1.50 diopters (D) (axis 90 +/- 15, 180 +/- 15) or -1.75 D (axis 90 +/- 10, 180 +/- 10)
* Adapted soft contact lens wearer
* Swims no more than once a week
* Has a wearable pair of spectacles.

Exclusion Criteria:

* Any ocular or systemic disorder which may contraindicate contact lens wear
* Any topical ocular medication
* Aphakic
* Corneal refractive surgery
* Corneal distortion from hard CL wear or keratoconus
* Pregnant or lactating
* Grade 2 or worse slit lamp signs
* Infectious disease
* Previous clinical study within 2 weeks
* Don't agree to participate
* Polymethyl methacrylate (PMMA) or rigid gas-permeable (RGP) lens wear in last 8 weeks
* Previous adverse effects that contraindicate extended lens wear.
* Self-reported symptoms of itchiness or scratchiness with habitual lenses.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2007-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Boston, Massachusetts, United States
- Australia (7):
  - Newtown, New South Wales
  - Camberwell, Victoria
  - Hawthorn, Victoria
  - Keilor, Victoria
  - Melbourne, Victoria
  - Mitcham, Victoria
  - Yallourn, Victoria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred at 1 site in the USA (n=50 enrolled), and 7 sites in Australia (n=62 enrolled)
Pre-assignment Details: Total of 112 subjects enrolled, 77 subjects completed study after 3 months. The study was then restricted down to two sites (Australia only) after 3 months with only 37 of the 77 being included. There were 36 subjects whom completed the full 6 month trial period.
Groups:
- Senofilcon A Bilaterally: Senofilcon A lenses worn daily bilaterally (in both eyes) for 3 months, replaced weekly. For those subject who continued the study from 3 months to 6 months, the same treatment was repeated.
- Balafilcon A Bilaterally: Balafilcon A lenses worn daily bilaterally (in both eyes) for 3 months, replaced weekly. For those subject who continued the study from 3 months to 6 months, the same treatment was repeated.
- Senofilcon A Toric/Balafilcon A Toric Contralaterally: Senofilcon A toric lens worn in one eye and Balafilcon A toric lens worn in the other eye (contralaterally), daily for 3 months, replaced weekly. For those subject who continued the study from 3 months to 6 months, the same treatment was repeated.
Period: Baseline to Month 3 (Period 1)
Arm/Group | Senofilcon A Bilaterally | Balafilcon A Bilaterally | Senofilcon A Toric/Balafilcon A Toric Contralaterally
Started | 36 | 25 | 51
Completed | 26 | 19 | 32
Not Completed | 10 | 6 | 19
Not completed — Adverse Event | 4 | 3 | 6
Not completed — Lost to Follow-up | 6 | 3 | 13
Period: Month 3 to Month 6 (Period 2)
Arm/Group | Senofilcon A Bilaterally | Balafilcon A Bilaterally | Senofilcon A Toric/Balafilcon A Toric Contralaterally
Started | 9 | 5 | 23
Completed | 9 | 4 | 23
Not Completed | 0 | 1 | 0
Not completed — Pregnancy | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Senofilcon A Toric Bilaterally | Balafilcon A Toric Bilaterally | Senofilcon A/Balafilcon A Contralaterally | Total
Number analyzed (Participants) | 36 | 25 | 51 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (6.9) | 30.4 (7.8) | 29.6 (8.6) | 29.8 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 19 | 35 | 79
  Male | 11 | 6 | 16 | 33
Region of Enrollment [Number; unit: participants]
  United States | 16 | 11 | 20 | 47
  Australia | 20 | 14 | 31 | 65

OUTCOME MEASURES:

1. Primary Outcome: Corneal Staining
Description: Scale of 0 to 4; 0=None, 1=Trace, 2=Mild, 3=Moderate, 4=Severe. The subjects were assigned to senofilcon A toric/balafilcon A toric contralaterally or senofilcon A or balafilcon A lenses bilaterally.
Time Frame: at 3 months of lens wear (period 1)
Population: Subjects analyzed included those who were enrolled, randomized to a study arm, and completed the study at 3 months, (n=77). Subjects were analyzed by device therefore the subjects from the contralateral arm were counted once in EITHER of the device arms for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Groups:
- Senofilcon A: Senofilcon A lenses worn daily bilaterally (in both eyes) for 3 months, replaced weekly. OR Senofilcon A Toric worn contralaterally, replaced weekly. (Due to the randomization and large number of non-completed it is possible that the contralateral subjects are not equally split between the devices.)
- Balafilcon A: Balafilcon A lenses worn daily bilaterally (in both eyes) for 3 months, replaced weekly OR Balafilcon A Toric worn contralaterally , replaced weekly. (Due to the randomization and large number of non-completed it is possible that the contralateral subjects are not equally split between the devices.)
Arm/Group | Senofilcon A | Balafilcon A
Number analyzed (Participants) | 42 | 35
Number analyzed (eyes) | 68 | 54
units on a scale | 0.6 (0.61) | 0.8 (0.74)

2. Primary Outcome: Limbal Redness
Description: as for outcome 1
Time Frame: at 3 months of lens wear (period 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Senofilcon A | Balafilcon A
Number analyzed (Participants) | 42 | 35
Number analyzed (eyes) | 68 | 54
units on a scale | 0.7 (0.61) | 0.7 (0.58)

3. Primary Outcome: Bulbar Redness
Description: as for outcome 1
Time Frame: at 3 months of lens wear (period 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Senofilcon A | Balafilcon A
Number analyzed (Participants) | 42 | 35
Number analyzed (eyes) | 68 | 54
units on a scale | 0.9 (0.58) | 0.8 (0.57)

4. Primary Outcome: Tarsal Roughness
Description: as for outcome 1
Time Frame: at 3 months of lens wear (period 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Senofilcon A | Balafilcon A
Number analyzed (Participants) | 42 | 35
Number analyzed (eyes) | 68 | 54
units on a scale | 1.1 (0.58) | 1.0 (0.75)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Senofilcon A: senofilcon A lenses (test) worn daily bilaterally (in both eyes) for 6 months, replaced weekly OR senofilcon A toric lenses worn contralaterally for 6 months, replaced weekly. All enrolled subjects are included. Subjects are counted by device, there are some subjects that are counted in both arms that are from the contralateral group, as identified in the participant flow.
- Balafilcon A: balafilcon A lenses (control) worn daily bilaterally (in both eyes) for 6months, replaced weekly OR balifilcon A toric lenses worn contralaterally for 6 months, replaced weekly. All enrolled subjects are included. Subjects are counted by device, there are some subjects that are counted in both arms that are from the contralateral group, as identified in the participant flow.
Arm/Group | Senofilcon A | Balafilcon A
Serious Adverse Events (participants affected / at risk) | 0/87 | 1/76
Other Adverse Events (participants affected / at risk) | 13/87 | 9/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Senofilcon A (N=87) | Balafilcon A (N=76)
Microbial Karatitis (Eye disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Senofilcon A (N=87) | Balafilcon A (N=76)
Non-Significant Events (Eye disorders) | 13 (13) | 9 (9) — These were reported non-specifically as a single category of non-significant events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication requires agreement and written consent from the Sponsor.